CLINICAL TRIAL: NCT00330915
Title: A Feasibility Study of Pemetrexed Single Agent and Folic Acid Given as Neoadjuvant Treatment in Patients With Resectable Rectal Cancer
Brief Title: A Study of Pemetrexed and Folic Acid Given Before Surgery (Neoadjuvant Treatment) to Patients With Rectal Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9732; H3E-MC-S077
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-06

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m2, intravenous (IV), every 21 days x 3 cycles
  Other Names: LY231514; Alimta

SUMMARY:
The purpose of this study is to help answer the following research questions:

If the study drug Pemetrexed can help patients with rectal cancer; If molecular biological parameters are correlated respectively changing due to cytotoxic treatment with Pemetrexed; To evaluate adverse events

ELIGIBILITY:
Inclusion Criteria:

* no prior therapy for rectal cancer
* pathological/ cytological diagnosis of adenocarcinoma of the rectum. Patients must have operable rectal cancer that is amenable to surgery.
* adequate organ function
* Eastern Cooperative Oncology Group (ECOG) Performance status 0 or 1
* signed informed consent
* at least 18 years of age
* surgically sterile, postmenopausal (women) or compliant with a medically approved contraceptive regimen during and for 6 months after the treatment.

Exclusion Criteria:

* concurrent administration of any other anti-tumor therapy
* treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* serious concomitant systemic disorders
* previously completed or withdrawn from this study
* pregnant or breast-feeding
* second primary malignancy
* history of significant neurological or mental disorder, including seizures or dementia
* inability to interrupt aspirin or other nonsteroidal anto-inflammatory drugs (NSAIDs)
* presence of clinically relevant third space fluid collections that cannot be controlled by drainage or other procedure prior to the study entry
* inability or unwillingness to take folic acid, vitamin B12 or dexamethasone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5PM Eastern time (UTC/ GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gothenburg, Sweden

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pemetrexed
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed
Number analyzed (Participants) | 37
Age Continuous [Mean (Standard Deviation); unit: years] | 60.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 26
Region of Enrollment [Number; unit: participants]
  Sweden | 37
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 37
    1 - Ambulatory, Restricted Strenuous Activity | 0
    2 - Ambulatory, No Work Activities | 0
    3 - Partially Confined to Bed, Limited Self Care | 0
    4 - Completely Disabled | 0
Histopathological Diagnosis [Number; unit: participants] — Assesses the extent to which cancer cells are similar in appearance and function to healthy cells of the same tissue type. Grades range from 1 (least aggressive and best prognosis) to 4 (most aggressive and worst prognosis).
  participants
    G1 - Well-Differentiated | 3
    G2 - Moderately Differentiated | 25
    G3 - Poorly Differentiated | 3
    Not Applicable | 4
    Unspecified | 2
Race/Ethnicity [Number; unit: participants]
  Caucasian | 36
  East Asian | 1
Blood Pressure [Mean (Standard Deviation); unit: mm Hg]
  Systolic Blood Pressure | 136.5 (18.4)
  Diastolic Blood Pressure | 77.6 (9.1)
Body Height [Mean (Standard Deviation); unit: centimeters] | 173.4 (9.4)
Body Surface Area [Mean (Standard Deviation); unit: meter squared] — BSA is derived as ((height[cm] x weight[kg])/3600)1/2
  meter squared | 2.0 (0.2)
Body Weight [Mean (Standard Deviation); unit: kilograms] | 80.4 (15.2)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 80.4 (14.8)
Time Since Initial Pathological Diagnosis [Mean (Standard Deviation); unit: weeks] — One patient is excluded because his pathological diagnosis occured 3.6 weeks after the date of informed consent.
  weeks | 3.2 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Pemetrexed Prior to Surgery
Description: Feasibility was defined as the ability to receive the total planned dose of Pemetrexed administered over a period of no more than 9 weeks permitting scheduling conflict. A ±5 percent variance in the calculated total dose was allowed.
Time Frame: 3 cycles (21-day cycles)
Population: Number of participants enrolled.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 37
participants
  Feasibility - Yes | 33
  Feasibility - No | 4

2. Secondary Outcome: Pathological Complete Response (pCR)
Description: Pathological complete response was defined as the absence of any tumor cells.
Time Frame: surgery following 3 cycles (21-day cycles) of chemotherapy
Population: Number of participants enrolled.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 37
participants
  Complete Response - Yes | 0
  Complete Response - No | 1
  Complete Response - Not Determined | 36

3. Secondary Outcome: Number of Participants With Complete Tumor Resection
Time Frame: surgery following 3 cycles (21-day cycles) of chemotherapy
Population: Number of participants enrolled.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 37
participants | 37

4. Secondary Outcome: Number of Participants Receiving Sphincter Saving Surgery
Time Frame: surgery following 3 cycles (21-day cycles) of chemotherapy
Population: Number of participants enrolled.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 37
participants
  Surgery - Yes | 25
  Surgery - No | 12

ADVERSE EVENTS:
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 17
Other Adverse Events (participants affected / at risk) | 37
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed
Atrial fibrillation (Cardiac disorders) | 1/37 (1)
Myocardial ischaemia (Cardiac disorders) | 1/37 (1)
Abdominal pain (Gastrointestinal disorders) | 1/37 (1)
Diarrhoea (Gastrointestinal disorders) | 2/37 (2)
Ileus (Gastrointestinal disorders) | 5/37 (5)
Vomiting (Gastrointestinal disorders) | 1/37 (1)
Pyrexia (General disorders) | 1/37 (1)
Anorectal infection (Infections and infestations) | 1/37 (1)
Infection (Infections and infestations) | 1/37 (1)
Peritoneal abscess (Infections and infestations) | 1/37 (1)
Pneumonia (Infections and infestations) | 1/37 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1/37 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1/37 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1/37 (1)
Wound complication (Injury, poisoning and procedural complications) | 3/37 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1/37 (1)
Haematoma (Vascular disorders) | 1/37 (1)
Haemorrhage (Vascular disorders) | 1/37 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed
Neutropenia (Blood and lymphatic system disorders) | 2/37 (2)
Lacrimation increased (Eye disorders) | 17/37 (18)
Abdominal pain (Gastrointestinal disorders) | 2/37 (2)
Constipation (Gastrointestinal disorders) | 2/37 (2)
Diarrhoea (Gastrointestinal disorders) | 7/37 (7)
Dry mouth (Gastrointestinal disorders) | 6/37 (6)
Dyspepsia (Gastrointestinal disorders) | 3/37 (3)
Frequent bowel movements (Gastrointestinal disorders) | 2/37 (2)
Nausea (Gastrointestinal disorders) | 18/37 (23)
Fatigue (General disorders) | 23/37 (33)
Mucosal inflammation (General disorders) | 4/37 (5)
Pain (General disorders) | 4/37 (5)
Pyrexia (General disorders) | 6/37 (7)
Alanine aminotransferase increased (Investigations) | 4/37 (4)
Haemoglobin decreased (Investigations) | 2/37 (6)
Neutrophil count decreased (Investigations) | 3/37 (5)
Weight decreased (Investigations) | 2/37 (2)
Anorexia (Metabolism and nutrition disorders) | 2/37 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 7/37 (7)
Dysgeusia (Nervous system disorders) | 2/37 (2)
Headache (Nervous system disorders) | 7/37 (7)
Pollakiuria (Renal and urinary disorders) | 2/37 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2/37 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2/37 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 9/37 (14)
Haemorrhage (Vascular disorders) | 2/37 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days